CLINICAL TRIAL: NCT02937220
Title: Influence of Superstructure Material on Crestal Bone Resorption and Esthetic Outcome of Dental Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Roshdy Radwan, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-10-223
Record Dates: First submitted 2016-10-16; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Single Tooth Dental Implant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monolithic zirconia crowns (Experimental): New crown material to restore dental implants
  Interventions: Procedure: monolithic zirconia crown
- metal ceramic crowns (Active Comparator): conventional crown material for restoring dental implants
  Interventions: Procedure: metal ceramic crown

INTERVENTIONS:
Procedure: monolithic zirconia crown — New crown material used as final restoration for dental implants
  Arms: Monolithic zirconia crowns
Procedure: metal ceramic crown — Conventional crown material used as final restoration for dental implants
  Arms: metal ceramic crowns

SUMMARY:
The aim of this study is to evaluate the influence of superstructure material on crestal bone resorption and esthetic outcome of dental implants in patients with single missing tooth in the aesthetic zone.

DETAILED DESCRIPTION:
The transfer of occlusal forces to the implant bone interface greatly influence the long term prognosis of implants and crestal bone resorption. Accordingly this study will investigate the influence of metal ceramic crowns and monolithic zirconia crowns on crestal bone resorption under loading. Also these crown materials greatly influence the final aesthetic outcome of the definitive restoration, which will be evaluated using the pink and white aesthetic scoring systems.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 18 years old.
2. Patients able to read and sign the informed consent document. 3. Medically free patients or with controlled systemic disease.

4. Patients with good bone quality and quantity evaluated using C.B.C.T. 5. Patients willing to return for follow-up examinations and evaluation. 6. Patients having single missing recently extracted premolar tooth.

Exclusion Criteria:

1. Young patients in growth stage.
2. Patients with unsuitable implantation sites (patients with major boney defects or sever bone resorption)
3. Pregnant women to avoid any complication that may occur in dental office.
4. Patients with uncontrolled systemic disease (hypertensive patient or uncontrolled diabetic patient)
5. Psychiatric problems or unrealistic expectations.
6. Multiple adjacent missing teeth.
7. Patients with bad oral hygiene

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
P.E.S. | 1 year
  Pink aesthetic scoring system for soft tissue aesthetics

SECONDARY OUTCOMES:
crestal bone resorption | 1 year

IPD SHARING:
Plan to Share IPD: Undecided